CLINICAL TRIAL: NCT05763836
Title: Comparison of the Analgesic Effects of Scalp Nerve Block and Intravenous Ibuprofen Applications Under the Guidance of Nociception Level Index (NoL) in Patients Undergoing Elective Supratentorial Craniotomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Ahmet Cem Ceran, Principal Investigator, Ankara University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: AU-AUFM-MECO.CERAN.ERKOC-23001
Record Dates: First submitted 2023-02-08; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Supratentorial Brain Tumor
Keywords: supratentorial craniotomy; scalp nerve block; intravenous ibuprofen; nociception level index; opioid reducing analgesia
MeSH Terms: interventions — Ibuprofen; Injections, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Block (Active Comparator): Scalp nerve block applied group
  Interventions: Procedure: Scalp nerve block
- Group Ibuprofen (Experimental): Intravenous ibuprofen applied group
  Interventions: Drug: Ibuprofen 800 Mg in 8 mL INTRAVENOUS INJECTION [Caldolor]
- Grup Ibuprofen&Block (Experimental): Both intravenous ibuprofen and scalp nerve block applied group
  Interventions: Drug: Ibuprofen 800 Mg in 8 mL INTRAVENOUS INJECTION [Caldolor]; Procedure: Scalp nerve block

INTERVENTIONS:
Drug: Ibuprofen 800 Mg in 8 mL INTRAVENOUS INJECTION [Caldolor] — Intravenous ibuprofen infusion
  Arms: Group Ibuprofen; Grup Ibuprofen&Block
Procedure: Scalp nerve block — Scalp nerves blocked by using local anesthetics
  Arms: Group Block; Grup Ibuprofen&Block

SUMMARY:
Introduction: Scalp incision is a powerful nociceptive stimulus that can exacerbate rapid changes in hemodynamic and sympathetic activity. Management of hemodynamic stability is essential in neuro-anesthesia and can be challenging among neurosurgery anesthesiologists. Neurosurgery operations include steps with a lot of painful stimuli such as intubation, insertion of a head-pinning, and craniotomy. A good anesthetic technique can improve hemodynamic responses by reducing the incidence of complications such as intracranial hypertension, bleeding, and longer recovery time. Routine analgesic approach in the intraoperative and postoperative period of supratentorial craniotomy includes the routine use of paracetamol, opioids, scalp nerve block with proven effectiveness, and intravenous ibuprofen, which gives good results by reducing opioid doses in moderate-to-severe pain. Supratentorial craniotomy surgery, which requires tight hemodynamic control, needs effective analgesic methods.

Trial design: It is a prospective, randomized controlled, consisting of factorial groups, double-blind study.

Participants: This study will be carried out at Ankara University Faculty of Medicine İbni Sina Hospital (Altındağ, Ankara, Turkey) between November 2022 and February 2023. One hundred and two ASA I-III patients with a body mass index (BMI) below 30, aged between 18 and 65, who will undergo elective supratentorial craniotomy due to a brain tumor, are planned to be included in the study.

Interventions: The group in which IV ipurofen was administered was named Ibuprofen Group (Group I), the group in which scalp nerve block was applied Block Group (Group), and the group in which IV ibuprofen and scalp nerve block were applied together was named Ibuprofen+Block Group (IB Group). In the premedication unit, 800 mg of ibuprofen in 100 ml of normal saline will be administered to Group I and Group IB, and 100 ml of normal saline without ibuprofen will be administered to Group B as a 30-minute IV infusion. After intubation, a scalp nerve block with 20 ml of 0.5% bupivacaine will be applied to Group B and Group IB, and 20 ml of normal saline will be injected into the block sites in Group I.

Objective: The investigators aimed to show the effect of scalp nerve block and IV ibuprofen applications, which are routinely applied, on the optimization of the patient's process from induction to the early postoperative period. In addition, the investigators will examine the comparison of hemodynamic and analgesic effects of scalp nerve block and IV ibuprofen applications under the guidance of pain monitor, and their contribution to reducing opioid consumption, which has side effects such as postoperative nausea/vomiting, slowing of GI motility, respiratory depression.

Outcome: The primary endpoint of the study was the differences between the groups in the changes in the patients' nociception level (NoL) index, heart rate, and blood pressure parameters at the time of head-pinning and the first surgical skin incision.

Randomization: Randomization of the patients into 3 groups will be carried out using the closed envelope method.

Blinding: The patients included in the study and the practicing anesthesiologist do not know which patient is included in which group.

DETAILED DESCRIPTION:
Scalp incision is a powerful nociceptive stimulus that can exacerbate rapid changes in hemodynamic and sympathetic activity. Management of hemodynamic stability is essential in neuro-anesthesia and can be challenging among neurosurgery anesthesiologists. A good anesthetic technique can improve hemodynamic responses by reducing the incidence of complications such as intracranial hypertension, bleeding, and longer recovery time. The stable hemodynamic not only provide an easy-to-perform surgical field, but also prevent serious complications such as bleeding, aneurysm rupture, and cerebral ischemia. In patients with impaired cerebral autoregulation, even a small increase in systemic arterial blood pressure can cause unexpected spikes in cerebral blood flow and intracranial pressure.

Neurosurgery operations include steps with a lot of painful stimuli such as intubation, insertion of a head-pinning, and craniotomy. In these patients where autoregulation may be impaired, it is extremely important to monitor the pain and provide adequate analgesia as well as providing sufficient depth of anesthesia in order to keep the hemodynamics stable.

Craniotomy consists of the steps of such as head-pinning in order to stabilize the head, making a skin incision, cutting the skull bone and removing the dura-mater and reaching the brain parenchyma. This process, which ends with the dura-mater incision, which the investigators define as the early intraoperative period, is the time period in which the most painful stimulus is observed, and accordingly, the increase in the level of vasoactive agents causes an increase in heart rate and blood pressure. In 86% of patients, there is pain of somatic origin, possibly involving soft tissue and pericranial muscles. Pain in this process is generally moderate to severe pain.

It has been reported that the pain after craniotomy is less than the pain after lumbar laminectomy for lumbar disc herniation. However, it has been shown that moderate-to-high pain may occur after craniotomy, especially in the first 2 hours postoperatively, and this is more common than previously thought. Increased oxygen consumption and catecholamine release caused by postoperative pain may predispose to intracranial hematomas by causing brain hyperemia and increased intracranial pressure. Local anesthetic infiltration or systemic analgesics such as non-steroidal anti-inflammatory drugs and opioids are used for craniotomy pain palliation. If the patient is conscious and feels pain after craniotomy, effective analgesia should be provided.

Routine analgesic approach in the intraoperative and postoperative period of supratentorial craniotomy includes the routine use of paracetamol, opioids, scalp nerve block with proven effectiveness, and intravenous (IV) ibuprofen, which gives good results by reducing opioid doses in moderate-to-severe pain. There are studies comparing drugs such as opioids, non-steroidal anti-inflammatory drugs (NSAIDs), ketamine, IV lidocaine, gabapentin in the prevention of the sympathetic response that occurs when entering the spiked cap and in the prevention of post-craniotomy pain and among these, scalp nerve block is accepted as the most effective analgesic approach.

Supratentorial craniotomy surgery, which requires tight hemodynamic control, needs effective analgesic methods. In this study, the investigators aimed to show the effect of scalp nerve block and IV ibuprofen applications, which are routinely applied, on the optimization of the patient's process from induction to the early postoperative period. In addition, the investigators will examine the comparison of hemodynamic and analgesic effects of scalp nerve block and IV ibuprofen applications under the guidance of pain monitor, and their contribution to reducing opioid consumption, which has side effects such as postoperative nausea/vomiting, slowing of GI motility, respiratory depression.

It is a prospective, randomized controlled, double-blind study. Randomization of the patients into 3 groups will be carried out using the closed envelope method. The group in which IV ipurofen was administered was named Ibuprofen Group (Group I), the group in which scalp nerve block was applied Block Group (Group), and the group in which IV ibuprofen and scalp nerve block were applied together was named Ibuprofen+Block Group (IB Group). The patients included in the study and the practicing anesthesiologist do not know which patient is included in which group.

Fentanyl (1-2 μg/kg) and propofol (2-3 mg/kg) will be used for anesthesia induction. Rocuronium (0.6 mg/kg) will be used as a muscle relaxant. Anesthesia maintenance will be provided with propofol and remifentanil infusion, keeping the bispectral index (BISTM) between 40-60 and the nociception level (NoL) index (PMD-200TM) between 10-25. The neuromuscular block depths of the patients will be monitored with train-of-four (TOF). As components of multimodal analgesia, 1 g paracetamol and 1.5 g magnesium sulfate will be administered as IV infusion to all patients after induction. Propofol and remifentanil infusions will be stopped after the end of the surgical procedure. Patients who have the appropriate level of consciousness and can perform simple commands will be extubated after the BIS value is above 80 and the TOF percentage is above 90.

In the premedication unit, 800 mg of ibuprofen in 100 ml of normal saline will be administered to Group I and Group IB, and 100 ml of normal saline without ibuprofen will be administered to Group B as a 30-minute IV infusion. After the infusion is over, the patients will be taken to the operating table. After the monitoring is completed, induction will be made and intubated.

After intubation, a scalp nerve block with 20 ml of 0.5% bupivacaine will be applied to Group B and Group IB, and 20 ml of normal saline will be injected into the block sites in Group I. Head stabilization will be achieved with a spiked head 5 minutes after the block application is completed. Normal saline solutions containing or not containing ibuprofen and the injectors used in the block will be prepared by the anesthesia technicians and the practicing anesthetist will be kept unaware of the content of the applied substance.

If the NoL value rises above 25 at all stages of the surgical process, an IV bolus of 0.5 mcg/kg remifentanil will be administered as a rescue analgesic.

Demographic characteristics such as the patient's name, surname, gender, age, weight, co-morbidities, American Society of Anesthesiologists (ASA) score will be recorded in the data collection form. In the intraoperative process, heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP), NoL value, BIS value parameters will be recorded before intubation, after intubation, before head-pinning, after head-pinning, before surgical incision, after surgical incision, before craniotomy, after craniotomy, before dura mater incision, and after dura mater incision.

In the intraoperative process, the times when rescue analgesics are needed will be recorded.

SPSS 11.5 program will be used in the analysis of the data. Mean±standard deviation and median (minimum-maximum) will be used for quantitative variables, and the number of patients (percentage) for qualitative variables. The Kruskal Wallis H test will be used to determine whether there is a difference between the categories of a qualitative variable with more than two categories in terms of quantitative variables, since the assumptions of normal distribution are not provided. Chi-square and Fisher exact tests will be used when the relationship between two qualitative variables is desired. To look at the before-after differences of the same measurement, if normal distribution assumptions are provided, the Paired-t test will be used, otherwise the Wilcoxon Sign test will be used. Statistical significance level will be taken as 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective suptatentorial craniotomy surgery
* Body Mass Index (BMI) below 30
* ASA I-III patient

Exclusion Criteria:

* Patients with a history of allergic reaction to the drugs to be used in the study
* Patients with heart, kidney and liver failure
* Patients who refused to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-05 (Estimated)

PRIMARY OUTCOMES:
Nociception level (NoL) index | From the beginning of the operation until the 3rd hour after the operation
  In this study, the difference between the groups in the change of NoL values due to the procedures applied in supratentorial craniotomy surgery will be evaluated. NoL values range between 0 and 100. Values above 25 indicate that the patient has pain, and the value increases as the pain increases.

SECONDARY OUTCOMES:
Heart rate | Heart rate measurements will be recorded during surgery.
  In this study, the difference between the groups in the change of heart rate due to the procedures applied in supratentorial craniotomy surgery will be evaluated. It will be evaluated as beat per minute.
Opioid consumption | After the induction of anesthesia, opioid infusion will be started and continued until the operation is completed and the maintenance of anesthesia is terminated. At the end of the surgery, the total amount of opioid consumed will be recorded.
  In the study, the amount of opioid consumed during surgery between groups will be compared. The amounts of remifentanil used as an opioid will be compared. The unit will be mcg.
Visual Analog Scale | 1st, 2nd and 3rd hours after surgery
  Patients will be asked to rate their pain status on a scale of 1 to 10 at 1, 2, and 3 hours after the end of surgery. Higher values indicate more pain.
Systolic blood pressure | Systolic blood pressure measurements will be recorded during surgery.
  In this study, the difference between the groups in the change of systolic blood pressure due to the procedures applied in supratentorial craniotomy surgery will be evaluated. The unit will be mmHg.
Dystolic blood pressure | Dystolic blood pressure measurements will be recorded during surgery.
  In this study, the difference between the groups in the change of dystolic blood pressure due to the procedures applied in supratentorial craniotomy surgery will be evaluated. The unit will be mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Başak Ceyda Meço, Study Director — Ankara University
Locations (1):
- Ankara University Fakulty of Medicine, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data collected to reach outcomes will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: For 1 year from the date of publication
Access Criteria: Academic institutions and individuals who have reached via e-mail

REFERENCES:
- [Background] Nemergut EC, Durieux ME, Missaghi NB, Himmelseher S. Pain management after craniotomy. Best Pract Res Clin Anaesthesiol. 2007 Dec;21(4):557-73. doi: 10.1016/j.bpa.2007.06.005. PMID 18286837
- [Background] Chen Y, Ni J, Li X, Zhou J, Chen G. Scalp block for postoperative pain after craniotomy: A meta-analysis of randomized control trials. Front Surg. 2022 Sep 26;9:1018511. doi: 10.3389/fsurg.2022.1018511. eCollection 2022. PMID 36225222
- [Background] Ban VS, Bhoja R, McDonagh DL. Multimodal analgesia for craniotomy. Curr Opin Anaesthesiol. 2019 Oct;32(5):592-599. doi: 10.1097/ACO.0000000000000766. PMID 31306155
- [Background] Vahabi S, Nadri S, Izadi F. The effects of gabapentin on severity of post spinal anesthesia headache. Pak J Pharm Sci. 2014 Sep;27(5):1203-7. PMID 25176361
- [Background] LASSEN NA. Cerebral blood flow and oxygen consumption in man. Physiol Rev. 1959 Apr;39(2):183-238. doi: 10.1152/physrev.1959.39.2.183. No abstract available. PMID 13645234
- [Background] Vahabi S, Rafieian Y, Abbas Zadeh A. The Effects of Intraoperative Esmolol Infusion on the Postoperative Pain and Hemodynamic Stability after Rhinoplasty. J Invest Surg. 2018 Apr;31(2):82-88. doi: 10.1080/08941939.2016.1278288. Epub 2017 Apr 4. PMID 28375035
- [Background] Hillman DR, Rung GW, Thompson WR, Davis NJ. The effect of bupivacaine scalp infiltration on the hemodynamic response to craniotomy under general anesthesia. Anesthesiology. 1987 Dec;67(6):1001-3. doi: 10.1097/00000542-198712000-00026. No abstract available. PMID 3318562
- [Background] Shiau JM, Chen TY, Tseng CC, Chang PJ, Tsai YC, Chang CL, Lee CG. Combination of bupivacaine scalp circuit infiltration with general anesthesia to control the hemodynamic response in craniotomy patients. Acta Anaesthesiol Sin. 1998 Dec;36(4):215-20. PMID 10399517
- [Background] Olsen KS, Pedersen CB, Madsen JB, Ravn LI, Schifter S. Vasoactive modulators during and after craniotomy: relation to postoperative hypertension. J Neurosurg Anesthesiol. 2002 Jul;14(3):171-9. doi: 10.1097/00008506-200207000-00001. PMID 12172288
- [Background] De Benedittis G, Lorenzetti A, Migliore M, Spagnoli D, Tiberio F, Villani RM. Postoperative pain in neurosurgery: a pilot study in brain surgery. Neurosurgery. 1996 Mar;38(3):466-9; discussion 469-70. doi: 10.1097/00006123-199603000-00008. PMID 8837797
- [Background] Vadivelu N, Kai AM, Tran D, Kodumudi G, Legler A, Ayrian E. Options for perioperative pain management in neurosurgery. J Pain Res. 2016 Feb 10;9:37-47. doi: 10.2147/JPR.S85782. eCollection 2016. PMID 26929661
- [Background] Dunbar PJ, Visco E, Lam AM. Craniotomy procedures are associated with less analgesic requirements than other surgical procedures. Anesth Analg. 1999 Feb;88(2):335-40. doi: 10.1097/00000539-199902000-00021. PMID 9972752
- [Background] Quiney N, Cooper R, Stoneham M, Walters F. Pain after craniotomy. A time for reappraisal? Br J Neurosurg. 1996 Jun;10(3):295-9. doi: 10.1080/02688699650040179. PMID 8799542
- [Background] Haldar R, Kaushal A, Gupta D, Srivastava S, Singh PK. Pain following craniotomy: reassessment of the available options. Biomed Res Int. 2015;2015:509164. doi: 10.1155/2015/509164. Epub 2015 Oct 1. PMID 26495298
- [Background] Hansen MS, Brennum J, Moltke FB, Dahl JB. Suboptimal pain treatment after craniotomy. Dan Med J. 2013 Feb;60(2):A4569. PMID 23461986
- [Background] Skutuliene J, Banevicius G, Bilskiene D, Macas A. The effect of scalp block or local wound infiltration versus systemic analgesia on post-craniotomy pain relief. Acta Neurochir (Wien). 2022 May;164(5):1375-1379. doi: 10.1007/s00701-021-04886-0. Epub 2021 Jun 28. PMID 34181084
- [Background] Graham AC, Reid MM, Andrews PJ. Perception of pain experienced and adequacy of analgesia following elective craniotomy. Anaesthesia. 1999 Aug;54(8):814-5. doi: 10.1046/j.1365-2044.1999.01046.x. No abstract available. PMID 10460707
- [Background] Verchere E, Grenier B, Mesli A, Siao D, Sesay M, Maurette P. Postoperative pain management after supratentorial craniotomy. J Neurosurg Anesthesiol. 2002 Apr;14(2):96-101. doi: 10.1097/00008506-200204000-00002. PMID 11907388